CLINICAL TRIAL: NCT04385836
Title: Trial of Alpha One Antitrypsin Inhalation in Treating Patient With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, mohamed mahmoud mohamed othman, assistant consultant gastroenterology, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-0520- 076-K-02-H
Record Dates: First submitted 2020-05-10; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- alpha one antitrypsin group (Active Comparator): - we will give 8 ml of intravenous alpha one antitrypsin (alpha1-proteinase inhibitor (AATD)Glassia 50 ml) add to 2cm of normal saline solution as nebulizer every 12 hours for 5 days
  Interventions: Drug: alpha one antitrypsin inhalation
- placebo group (Placebo Comparator): we will give 8 ml of normal saline as nebulizer every 12 hours for 5 days
  Interventions: Drug: alpha one antitrypsin inhalation

INTERVENTIONS:
Drug: alpha one antitrypsin inhalation — - we will give 8 ml of intravenous alpha one antitrypsin (alpha1-proteinase inhibitor (AATD)Glassia 50 ml) as nebulizer every 12 hours for 5 days

SUMMARY:
It is clear now that SARS-CoV-2 could use angiotensin-converting enzyme 2 (ACE2), the same receptor as SARS-CoV Transmembrane protease serine type 2 (TMPRSS2), a protease belonging to the type II transmembrane serine protease family, cleaves the coronavirus spike protein Serine proteases are inhibited by a diverse group of inhibitors, The best-studied serpins are antithrombin and alpha 1-antitrypsin

ELIGIBILITY:
Inclusion Criteria:

1. Positive RT-PCR) assay for SARS-CoV-2
2. Age >18 years
3. Hospitalized
4. Able to give informed consent

Exclusion Criteria:

1. Known allergy to AAT
2. imminent death within next 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
clinical improvement | we will follow the patient daily starting from the day 0 which is the first day of giving drug for 3 weeks or till clinical improvement and discharge from the hospital or till death whichever comes first.
  Time to clinical improvement, from the point of randomization to two-point improvement on a seven-point ordinal scale or discharged alive from hospital, whichever comes first.
  Ordinal Scale - 1, Ambulatory with normal activities; 2, Ambulatory with limitation of normal activities; 3, not requiring supplemental oxygen; 4, requiring supplemental oxygen by mask or nasal prongs; 5, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6, requiring ECMO, invasive mechanical ventilation, or both; and 7, death

CONTACTS AND LOCATIONS:
Overall Officials: mohammed m othman, Principal Investigator — MOH
Locations (1):
- Ministry of Health, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes